CLINICAL TRIAL: NCT03243721
Title: Impact of Gilenya on Cognitive Function and Thalamic Volume Measured by 7 Tesla MRI in Multiple Sclerosis
Brief Title: Gilenya's Impact on Cognitive Function and Thalamic Volumes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Devon Conway MD, Principal Investigator, The Cleveland Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CCF 17-766
Record Dates: First submitted 2017-08-01; First posted 2017-08-09 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; thalamus; high field MRI; cognition
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: There will be two groups running in parallel. One will be MS patients (15) and the other will be control patients (5). Both groups will receive the same interventions.
Masking Description: There is no masking in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gilenya treated MS patients (Experimental): Multiple sclerosis patients treated with Gilenya for at least six months. This group will receive diagnostic tests: 7T MRI and Neurocognitive testing.
  Interventions: Diagnostic Test: 7T MRI; Diagnostic Test: Neurocognitive testing
- Healthy controls (Experimental): Subjects without multiple sclerosis or other diseases of the central nervous system. This group will receive diagnostic tests: 7T MRI and Neurocognitive testing.
  Interventions: Diagnostic Test: 7T MRI; Diagnostic Test: Neurocognitive testing

INTERVENTIONS:
Diagnostic Test: 7T MRI — A high field MRI that will take approximately one hour.
Diagnostic Test: Neurocognitive testing — A series of tests to assess memory, verbal skills, and visuospatial skills.

SUMMARY:
This evaluation will be a one-year feasibility study to characterize the neuroprotective benefits of Gilenya and its effects on cognition and grey matter volumes. The study will enroll 15 patients with relapsing-remitting multiple sclerosis being treated with Gilenya and 5 healthy controls. Each participant will undergo a battery of neurometric testing at baseline, six months, and one year. In addition, patients will undergo high-field 7T MRI at the same time points.

DETAILED DESCRIPTION:
Cognitive impairment is a well-recognized manifestation of multiple sclerosis (MS) with prevalence estimates ranging from 43 to 70%. It is also known to occur as early as the first demyelinating event and is a major factor contributing to quality of life in MS. Treatment strategies for cognitive impairment in MS are limited. Several agents have been tested as therapeutics for MS-related cognitive dysfunction and have showed no major benefit. Cognitive rehabilitation has shown some promise, but the data are limited and many studies have suffered from methodological shortcomings. Given the lack of well-established treatment options and the substantial impact of cognitive impairment, protection of cognitive function from the earliest stages of the disease is of great importance.

Cognitive outcomes received relatively little attention in the pivotal studies of MS disease modifying therapies (DMT), but some data suggest that DMT may have a positive impact on cognition. Gilenya is of special interest because it was found to have a significant protective effect on whole brain atrophy when compared against placebo and intramuscular interferon β-1a in two phase III studies, showing a 31-35% reduction in percentage brain volume change. Gilenya's effect on whole brain atrophy leads to the natural hypothesis that it may have a beneficial effect on cognitive function in MS. Also of particular interest is the extent to which protection of the thalamus and cortex contributes to Gilenya's effect on whole brain atrophy and possible effects on cognition.

The study will enroll 15 subjects from the Cleveland Clinic Mellen Center patient population. Participants must have been on Gilenya for at least 6 months at the time of study entry. The study will involve three assessments: at baseline, six months, and one year. At each time point, participants will undergo 7T MRI of the brain with and without contrast. Participants will also undergo a battery of neurometric testing at each time point. The tests will include the Brief Visuospatial Memory Test - Revised (visuospatial skills), the iPadTM Processing Speed Test (processing speed), the Selective Reminding Test (verbal learning and memory), and the Delis-Kaplan Executive Function System Sorting Test (problem-solving skills; can only be administered at baseline and one year due to version limitations).

ELIGIBILITY:
Inclusion Criteria (MS Patients):

1. RRMS phenotype
2. Treated with Gilenya for ≥6 months at the time of the baseline visit.
3. Age 18-50 inclusive.
4. EDSS 0-4.0
5. Disease duration of 5-15 years.
6. At least 12 years of education (high school diploma or general equivalency diploma).
7. Physically capable of completing neurometric testing and MRI studies.

Inclusion Criteria (Healthy Controls):

1. Age 18-50 inclusive.
2. At least 12 years of education (high school diploma or general equivalency diploma)
3. Physically capable of completing neurometric testing and MRI studies.

Exclusion Criteria (MS Patients):

1. Contraindication to MRI (e.g. metal implants)
2. Current use of immunomodulatory or immunosuppressant medications other than Gilenya.
3. Disease of the central nervous system other than MS (e.g. Alzheimer disease, stroke, epilepsy).
4. Use of anti-psychotic or psychostimulant medications. Patients started on modafinil or armodafinil more than six months prior to enrollment will not be excluded.
5. Ongoing major depressive disorder that, in the opinion of the investigator, may affect cognitive functioning.
6. MS relapse within 90 days of study entry.
7. Treatment with corticosteroids within 90 days of study entry.
8. Current illicit substance use.
9. History of alcohol or drug abuse.

Exclusion Criteria (Healthy Controls):

1. Contraindication to MRI (e.g. metal implants, claustrophobia).
2. Disease of the central nervous system (e.g. MS, Alzheimer disease, stroke, epilepsy).
3. Use of anti-psychotic or psychostimulant medications. Patients started on modafinil or armodafinil more than six months ago will not be excluded.
4. Ongoing major depressive disorder that, in the opinion of the investigator, may affect cognitive functioning.
5. Current illicit substance use.
6. History of alcohol or drug abuse.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
Thalamic volume to cognitive performance | One year.
  Spearman's correlation coefficient of change in thalamic volume and change in cognitive function from baseline to one year in RRMS patients treated with Gilenya.

SECONDARY OUTCOMES:
Thalamic volume to other MRI metrics | Six months and one year.
  Ratio of change in thalamic volume from baseline to six months and from baseline to one year to 1) change in brain volume (from baseline to six months and from baseline to one year); 2) change in T2 lesion volume (from baseline to six months and from baseline to one year); and 3) change in cortical thickness (from baseline to six months and from baseline to one year).
Thalamic nuclei to cognitive performance | Six months and one year.
  Spearman correlation coefficient for change in the volume of each thalamic nuclei (from baseline to six months and from baseline to one year) and change in cognitive testing scores (from baseline to six months and from baseline to one year).
Thalamic myelin density to cognitive performance | Six months and one year.
  Spearman correlation coefficient of change in thalamic myelin density (from baseline to six months and from baseline to one year) to change in cognitive test performance (from baseline to six months and from baseline to one year).
Thalamic axon density to cognitive performance | Six months and one year.
  Spearman correlation coefficient of change in thalamic axon density (from baseline to six months and from baseline to one year) to change in cognitive test performance (from baseline to six months and from baseline to one year).
Changes in MRI metrics in Gilenya treated patients vs. controls | Six months and one year.
  Ratio of change in each of the following between Gilenya treated MS patients and healthy controls: 1.) Thalamic volume change (from baseline to six months and from baseline to one year); 2) Cortical thickness change (from baseline to six months and from baseline to one year); 3) thalamic axon density change (from baseline to six months and from baseline to one year); 4) thalamic myelin density (from baseline to six months and from baseline to one year).
Changes in cognitive performance in Gilenya treated patients vs controls | Six months and one year.
  Ratio of change in cognitive test performance (from baseline to six months and from baseline to one year) between Gilenya treated patients and controls.
Thalamic volume to cognitive performance | Six months.
  Spearman's correlation coefficient of change in thalamic volume and change in cognitive function from baseline to six months in RRMS patients treated with Gilenya.

CONTACTS AND LOCATIONS:
Overall Officials: Devon S Conway, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
The data will be analyzed in aggregate. There is no plan to share individual participant data with other researchers.